CLINICAL TRIAL: NCT06347471
Title: The Transmission of Artemisinin Resistant Parasites Before and After Conventional Artemisinin-combination Therapy: a Longitudinal Study
Brief Title: The Transmission of Artemisinin Resistant Parasites Before and After Conventional Artemisinin-combination Therapy
Acronym: SPARTAN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Infectious Diseases Research Collaboration, Uganda (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBS-2023-477
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-03

CONDITIONS: Falciparum; Malaria
Keywords: Malaria Transmission; Artemisinin resistance; Gametocytes; Spread of resistance
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- artemether-lumefantrine (Active Comparator): artemether-lumefantrine according to manufacturer instructions
  Interventions: Drug: Artemether-lumefantrine
- dihydroartemisinin-piperaquine (Experimental): dihydroartemisinin-piperaquine according to manufacturer instructions
  Interventions: Drug: Dihydroartemisinin-Piperaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Participants in the Artemether-Lumefantrine arm will be treated with standard doses of AL (Coartem, Novartis). Tablets containing 20/80 mg artemether and 120/480 mg lumefantrine will be administered per manufacturer guidelines. All doses will be given under direct supervision with fatty food.
  Other Names: Coartem
  Arms: artemether-lumefantrine
Drug: Dihydroartemisinin-Piperaquine — Participants in the DHA-PPQ arm will be treated with standard doses of DHA-PPQ. Tablets containing 40 mg dihydroartemisinin/320 mg piperaquine tablets (Eurartesim, Sigma Tau or Duocotecxin, Beijing Holley-Cotect Pharmaceutical Co) will be administered per manufacturer guidelines. All doses will be given under direct supervision on an empty stomach, as per manufacturer instructions.
  Other Names: Eurartesim; Duocotecxin
  Arms: dihydroartemisinin-piperaquine

SUMMARY:
A prospective study will be carried out in an area where parasites with reduced sensitivity to malaria drugs (artemisinins) have recently emerged. The study will recruit participants from patients who attend the clinic with uncomplicated malaria and asymptomatically infected individuals. Participants are treated with conventional artemisinin-combination therapies (ACT) as part of standard clinical care. From this population, we will select P. falciparum gametocyte carriers.

Before, during and after ACT treatment, the transmission potential of artemisinin resistant and wild type infections will be assessed by microscopy, molecular methods, parasite culture and mosquito feeding assays. Parasite clearance will be determined in the first days (d0-3) after treatment.

The study population will consist of passively recruited patients with uncomplicated P. falciparum malaria and asymptomatically infected individuals who are microscopy positive for gametocytes. Participants will be treated with conventional therapies for uncomplicated malaria without randomization: artemether-lumefantrine (AL) or dihydroartemisinin-piperaquine (DHA-PPQ). All doses are supervised. Parasite clearance is assessed ex vivo by ring-stage survival assays and by daily slides during the first days of treatment.

Gametocyte carriage and gametocyte commitment/production will be determined for resistant and wild type infections before, during and after treatment. In addition, venous blood will be collected at three timepoints to assess transmission to mosquitoes before (d0), during (d2) and after treatment (d7). The total duration of participation will be 7 days, the primary endpoint will be the reduction in mosquito infection rates at d2 (artemether-lumefantrine) or d7 (dihydroartemisinin-piperaquine) compared to pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥2 years
* blood smear positive for P. falciparum gametocytes
* mono-infection with P. falciparum confirmed by positive blood smear;
* parasitaemia of >100 P. falciparum asexual forms/µL;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule;
* informed consent from parent or guardian;
* haemoglobin ≥ 7.0 g/dl for children below 10 years of age or ≥8.0g/dL for older individuals

Exclusion Criteria:

* presence of general danger signs;
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe malnutrition defined as a very low weight for height (below -3z scores of the median WHO growth standards), by visible severe wasting, or by the presence of nutritional oedema.
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean within person percent change (presented as percent reduction) in mosquito infection rate in infectious individuals from baseline. | day 2 vs day 0 (AL arm) and day 7 vs day 0 (DP arm)
  Mean within person percent change (presented as percent reduction) in mosquito infection rate in infectious individuals from baseline (day 0, pre-treatment) to day 2 post treatment in the AL and day 7 post-treatment in the DHA-PPQ arm. Infectivity is assessed by mosquito membrane feeding assays; percent reduction is calculated separately for ΔPfK13 vs wild type infections.

SECONDARY OUTCOMES:
Mean within person percent change (presented as percent reduction) in mosquito infection rate from baseline | days 0, 2, 7
  Mean within person percent change (presented as percent reduction) in mosquito infection rate from baseline to all feeding time-points. Infectivity is assessed by mosquito membrane feeding assays; comparisons are performed within treatment arms for ΔPfK13 vs wild type infections.
Mean oocyst intensity (in all/all infected mosquitoes) | days 0, 2, 7
  Mean oocyst intensity (in all/all infected mosquitoes) will be assessed at all feeding time-points; comparisons are performed within treatment arms for ΔPfK13 vs wild type infections
Male and female gametocyte sex ratio (proportion male) | days 0, 1, 2, 3, 7
  Male and female gametocyte sex ratio (proportion male) at all time-points, determined by molecular assays; comparisons are performed within treatment arms for ΔPfK13 vs wild type infections.
Gametocyte circulation time | days 0, 1, 2, 3, 7
  Gametocyte circulation time (cumulative), determined by microscopy or molecular assays, compared between treatment arms and between ΔPfK13 vs wild type infections
Gametocyte area under the curve | days 0, 1, 2, 3, 7
  Gametocyte area under the curve (cumulative), determined by microscopy or molecular assays, compared between treatment arms, and between ΔPfK13 vs wild type infections
Asexual parasite prevalence | days 0, 1, 2, 3, 7
  Asexual parasite prevalence at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms, between arms, and between ΔPfK13 vs wild type infections
Asexual parasite density | days 0, 1, 2, 3, 7
  Asexual parasite density at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms, between arms, and between ΔPfK13 vs wild type infections
Total parasite prevalence | days 0, 1, 2, 3, 7
  Total parasite prevalence at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms, between arms, and between ΔPfK13 vs wild type infections
Total parasite density | days 0, 1, 2, 3, 7
  Total parasite density at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms, between arms, and between ΔPfK13 vs wild type infections
The density of ΔPfK13 vs wild type genotypes | days 0, 1, 2, 3, 7
  The density of ΔPfK13 vs wild type genotypes in peripheral blood, the asexual parasite fraction and gametocyte fraction before and after initiation of treatment. The relative abundance of ΔPfK13 genotypes will be compared between pre- and post-treatment timepoints
The density of ΔPfK13 vs wild type genotypes in oocysts and sporozoites in mosquitoes that become infected before and after initiation of treatment | days 0, 2, 7
  The density of ΔPfK13 vs wild type genotypes in oocysts and sporozoites in mosquitoes that become infected before and after initiation of treatment. The relative abundance of ΔPfK13 genotypes will be compared between pre- and post-treatment timepoints
Mean within person percent change (presented as percent reduction) in mosquito infection rate from baseline after gametocyte enrichment | days 0, 2, 7
  Mean within person percent change (presented as percent reduction) in mosquito infection rate from baseline to all feeding time-points. Infectivity is assessed by mosquito membrane feeding assays after gametocyte enrichment; comparisons are performed within treatment arms for ΔPfK13 vs wild type infections.

CONTACTS AND LOCATIONS:
Overall Officials: Teun Bousema, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Uganda (2):
  - Dr. Ambrosoli Memorial Hospital, Kalongo, Agago district
  - Patongo Health Facility IV, Patongo, Agago district

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared through an online repository
Supporting Information: Study Protocol
Time Frame: Upon publication

REFERENCES:
- [Background] Conrad MD, Asua V, Garg S, Giesbrecht D, Niare K, Smith S, Namuganga JF, Katairo T, Legac J, Crudale RM, Tumwebaze PK, Nsobya SL, Cooper RA, Kamya MR, Dorsey G, Bailey JA, Rosenthal PJ. Evolution of Partial Resistance to Artemisinins in Malaria Parasites in Uganda. N Engl J Med. 2023 Aug 24;389(8):722-732. doi: 10.1056/NEJMoa2211803. PMID 37611122
- [Background] Tumwebaze PK, Conrad MD, Okitwi M, Orena S, Byaruhanga O, Katairo T, Legac J, Garg S, Giesbrecht D, Smith SR, Ceja FG, Nsobya SL, Bailey JA, Cooper RA, Rosenthal PJ. Decreased susceptibility of Plasmodium falciparum to both dihydroartemisinin and lumefantrine in northern Uganda. Nat Commun. 2022 Oct 26;13(1):6353. doi: 10.1038/s41467-022-33873-x. PMID 36289202